CLINICAL TRIAL: NCT02140216
Title: Allogeneic Red Cell Transfusion and Its Influence on Relevant Humoral and Cellular Immunological Parameters
Brief Title: Immunomodulation Effect of Blood Transfusion
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: Wolf Schleinzer Stiftung zur Wissenschafts- und Bildungsförderung, Germany (Unknown)
Responsible Party: Principal Investigator, Benno von Bormann, Professor, Mahidol University
Other Study IDs: Si 081/2557 (EC3)
Record Dates: First submitted 2014-05-05; First posted 2014-05-16 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Incompatible Blood Transfusion; Immune Defect; Surgery
Keywords: Blood transfusion; Immune; Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Day 0 blood transfusion: Patients undergoing elective spine surgery receiving intra- or immediate-postoperative red cell blood transfusion.
  Interventions: Biological: Day 0 blood transfusion
- Day 1 or 2 blood transfusion: Patients undergoing elective spine surgery receiving first red cell blood transfusion on day 1 or 2 after surgery.
  Interventions: Biological: Day 1 or 2 blood transfusion
- No blood transfusion: Patients undergoing elective spine surgery receiving no blood transfusion.
  Interventions: Biological: No blood transfusion

INTERVENTIONS:
Biological: No blood transfusion — No blood transfusion
  Groups: No blood transfusion
Biological: Day 0 blood transfusion — Patients undergoing elective spine surgery receiving intra- or immediate-postoperative red cell blood transfusion.
  Groups: Day 0 blood transfusion
Biological: Day 1 or 2 blood transfusion — Patients undergoing elective spine surgery receiving first red cell blood transfusion on day 1 or 2 after surgery.
  Groups: Day 1 or 2 blood transfusion

SUMMARY:
An increasing number of publications have demonstrated that homologous (allogeneic) blood transfusion impairs outcome in cancer and non-cancer patients. Leukocyte depletion of blood products cannot solve these problems, despite improved quality of red cells; a recent study demonstrated deteriorated outcome of cancer patients with elective colon surgery and transfusion of leukocyte depleted allogeneic blood.

DETAILED DESCRIPTION:
All patients undergo the identical anesthesiological procedure, including premedication, general anesthesia with endotracheal intubation, monitoring and postoperative pain therapy and mobilization.Surgery is performed by the identical team performing a standardized technique.

Transfusion regimen The 'trigger' for homologous red cell transfusion intra- and postoperatively is the actual hematocrit concentration. Transfusion depends on discretion of the treating physicians. Number of units transfused, amount of blood loss, time, reasoning and decision maker are recorded.

Blood samples Within the kind of surgical procedures chosen for this study the chance of red cell transfusion is about 60 - 70%. In terms of figures 10 non-transfused cases could be gained within 40 cases in total. However, transfusion or non-transfusion does not happen in a row. We expect the total number of patients with blood withdrawal to be between 50 and 60. Additionally withdrawn samples currently not used for analysis will stored for further studies.

The purpose to include non-transfused otherwise fully comparable patients is to distinguish between trauma (operation) and transfusion and their influence on immune modulation. Within the studies about blood transfusion and immune modulation only some few made this differentiation. In patients with colorectal cancer surgery randomized groups with autologous predonation and patients with allogeneic transfusion only have been compared. However, within the latter (allogeneic) group of 27 patients only 13 had to be transfused, thus creating a non-transfusion group of 14 patients. These 14 non-transfused patients remained within the study being compared with autologous and allogeneic transfused patients. Operative trauma and allogeneic transfusion both increased the secretion of several cytokines including tumor necrosis factor (TNF) alpha and Interleukin-10; this effect was less pronounced in patients with autologous- and without any transfusion. Another group studied forty three orthopedic patients with total knee- or hip-arthroplasty, initially to compare autologous to allogeneic red cell transfusion. They had to change their protocol due to the small number of allogeneic transfusions (8 of 43). Including perioperatively transfused patients only (n = 37) they found an increase in immune regulatory cytokine Interleukin (IL)-10 after red cell transfusion, which was most pronounced 7 days after surgery, whereas there was only a mild increase in non- or autologous transfused patients. Unfortunately they did not differentiate between autologous-and non-transfused patients. Thus their data could not reveal the effect of surgery itself on the analyzed parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective spine surgery
* American Society of Anesthesiologist Risk score classification (ASA) I-III
* Hemoglobin > 9 gm/dL

Exclusion Criteria:

* Patients who have the concomitant condition; cancer, history of heart disease including, heart failure, coronary artery disease, hypertension treated with more than one medicament, serum creatinine > 1.5 mg/dL., stroke, neurologic and mental deficits, epilepsy, general or local infection (site of surgery), coagulation disorders, rheumatoid arthritis.
* Patients who have one of the following drugs; aspirin, methotrexate, cyclosporin, qualaquin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective spine surgery/
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-06-18 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Macrophage inflammatory protein 1 alpha (MIP-1a) | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
macrophage inflammatoryprotein 1 beta (MIP-1b) | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
platelet-derived growth factor-BB | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
RANTES | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
tumour TNF alpha | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
VEGF | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
Ferritin | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
Fibrinogen | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
procalcitonin | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
interleukin | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
basic fibroblast growth factor (B-FGF) | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
eotaxin (monocyte chemotactic proteins) | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
G-CSF | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
GM-CSF | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
IFN-alpha | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
IP-10 | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
MCP-1 | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
MCAF | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
serum amyloid A | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
tissue plasminogen activator | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
Postoperative non-surgical complications | 30 days
  Infection, thrombosis, pulmonary affection

SECONDARY OUTCOMES:
CD2 Cellular immunologic parameter (non-radioisotope), | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
CD3 Cellular immunologic parameter (non-radioisotope), | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
CD4 Cellular immunologic parameter (non-radioisotope), | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
CD 8 Cellular immunologic parameter (non-radioisotope), | 5 days
  preoperative, postoperative day 1, 3, 5
CD 8 Cellular immunologic parameter (non-radioisotope), | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
CD 25 Cellular immunologic parameter (non-radioisotope), | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
CD 30 Cellular immunologic parameter (non-radioisotope), | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
CD 19 Cellular immunologic parameter (non-radioisotope), | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
CD 20 Cellular immunologic parameter (non-radioisotope), | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
CD 138 Cellular immunologic parameter (non-radioisotope), | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
CD 56 Cellular immunologic parameter (non-radioisotope), | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
CD 303 Cellular immunologic parameter (non-radioisotope), | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
CLT cytotoxicity (non-radioisotope), | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
CD 304 | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5
NK cytotoxicity | 5 days
  Blood sample on preoperative, postoperative day 1, 3, 5

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Study Director — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Background] Marik PE, Corwin HL. Efficacy of red blood cell transfusion in the critically ill: a systematic review of the literature. Crit Care Med. 2008 Sep;36(9):2667-74. doi: 10.1097/CCM.0b013e3181844677. PMID 18679112
- [Background] von Bormann B, Wirtz S, Weiler J, von Bormann C, Trobisch H. [Quality of whole blood as a result of storage and preparation (inline-leukocyte depletion). Evidence for autologous predeposit]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2000 May;35(5):326-32. doi: 10.1055/s-2000-323. German. PMID 10858843
- [Background] Ghio M, Contini P, Negrini S, Mazzei C, Zocchi MR, Poggi A. Down regulation of human natural killer cell-mediated cytolysis induced by blood transfusion: role of transforming growth factor-beta(1), soluble Fas ligand, and soluble Class I human leukocyte antigen. Transfusion. 2011 Jul;51(7):1567-73. doi: 10.1111/j.1537-2995.2010.03000.x. Epub 2011 Jan 7. PMID 21214580
- [Background] Leal-Noval SR, Munoz-Gomez M, Arellano V, Adsuar A, Jimenez-Sanchez M, Corcia Y, Leal M. Influence of red blood cell transfusion on CD4+ T-helper cells immune response in patients undergoing cardiac surgery. J Surg Res. 2010 Nov;164(1):43-9. doi: 10.1016/j.jss.2009.03.010. Epub 2009 Apr 18. PMID 19592026
- [Background] Heiss MM, Fasol-Merten K, Allgayer H, Strohlein MA, Tarabichi A, Wallner S, Eissner HI, Jauch KW, Schildberg FW. Influence of autologous blood transfusion on natural killer and lymphokine-activated killer cell activities in cancer surgery. Vox Sang. 1997;73(4):237-45. doi: 10.1046/j.1423-0410.1997.7340237.x. PMID 9407641
- [Derived] Suksompong S, Tassaneetrithep B, Ariyawatkul T, Sirivanasandha B, Wilartratsami S, Wongsa A, von Bormann B. Allogeneic red cell transfusion and its influence on relevant humoral and cellular immunological parameters: A prospective observational trial. Eur J Anaesthesiol. 2019 Nov;36(11):814-824. doi: 10.1097/EJA.0000000000001027. PMID 31157653